CLINICAL TRIAL: NCT04196803
Title: Methylomic Biomarkers, Magnesium Deficiency and Colon Neoplasia Prevention
Brief Title: Ancillary Study of Methylation Biomarkers in a Randomized Controlled Trial of a Personalized Prevention of Colorectal Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Qi Dai, Professor of Medicine, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 100106c; R01CA149633 (NIH); R01CA202936 (NIH); R01DK110166 (NIH)
Record Dates: First submitted 2019-12-10; First posted 2019-12-12 (Actual); Results first posted 2024-06-25 (Actual); Last update posted 2024-06-25 (Actual); Status verified 2024-06

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — magnesium diglycinate

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- magnesium treatment (Active Comparator): Participants were assigned to magnesium glycinate
  Interventions: Dietary Supplement: Magnesium glycinate
- placebo (Placebo Comparator): Participants were assigned to placebo group
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Magnesium glycinate — Oral administration of magnesium glycinate daily for 12 weeks
  Arms: magnesium treatment
Dietary Supplement: Placebo — Oral administration of identical-appearing placebo daily for 12 weeks
  Arms: placebo

SUMMARY:
Based on the magnesium tolerance test (MTT, "gold standard" for assessing magnesium (Mg) status), it was found that over 50% of participants in the US exhibited Mg deficiency. Studies suggest that the relationship between high Mg intake and disease risks may be varied by an individual's Mg status. Despite its importance, MTT is not commonly employed in routine clinical practice or research studies. Instead, serum Mg levels are typically used for clinical diagnosis, although this method has shown limited efficacy in identifying Mg deficiency accurately. Consequently, there is a pressing need to develop practical, sensitive, and specific biomarkers that can efficiently identify individuals with Mg deficiency.

It is known that DNA methylation changes are inducible by environmental exposures, including nutrients, and reversible when the exposure disappears. There are two major types of DNA methylation modifications, 5-hydroxymethylcytosine (5-hmC) and 5-methylcytosine (5-mC). 5-mC is often associated with suppressed gene expression. 5-hmC, generated by the oxidation of 5-mC, is specifically enriched in expressed genes and play a critical role in activating and/or maintaining gene expression. We plan identify 5-hmC and 5-mC for Mg deficiency by a 4- phase comprehensive epigenome-wide association study (EWAS) using the samples collected in the "Personalized Prevention of Colorectal Cancer Trial [PPCCT, R01CA149633; PI, Dai & Yu]" .

The parent trial [NCT04196023] that supports this ancillary research is a randomized controlled trial to evaluate the efficacy of reducing the Ca:Mg ratio among those who consume high Ca:Mg ratio diets to decrease the risk of colorectal cancer. For this ancillary trial research, the investigators are examining ancillary measures of Changes of Cytosine Modification in TMPRSS2.

ELIGIBILITY:
Inclusion Criteria:

1. Participants from our parent study (Personalized Prevention of Colorectal Cancer Trial, NCT#01105169, IRB#100106);
2. Participants consent to store/share biospecimens for future research.

Exclusion Criteria:

1. Participants cannot provide their blood samples in the parent study.

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2011-03-11 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

REFERENCES:
- [Background] Fan L, Zhu X, Zheng Y, Zhang W, Seidner DL, Ness R, Murff HJ, Yu C, Huang X, Shrubsole MJ, Hou L, Dai Q. Magnesium treatment on methylation changes of transmembrane serine protease 2 (TMPRSS2). Nutrition. 2021 Sep;89:111340. doi: 10.1016/j.nut.2021.111340. Epub 2021 May 7. PMID 34116393
- [Background] Fan L, Zhu X, Rosanoff A, Costello RB, Yu C, Ness R, Seidner DL, Murff HJ, Roumie CL, Shrubsole MJ, Dai Q. Magnesium Depletion Score (MDS) Predicts Risk of Systemic Inflammation and Cardiovascular Mortality among US Adults. J Nutr. 2021 Aug 7;151(8):2226-2235. doi: 10.1093/jn/nxab138. PMID 34038556
- [Background] Zhu X, Borenstein AR, Zheng Y, Zhang W, Seidner DL, Ness R, Murff HJ, Li B, Shrubsole MJ, Yu C, Hou L, Dai Q. Ca:Mg Ratio, APOE Cytosine Modifications, and Cognitive Function: Results from a Randomized Trial. J Alzheimers Dis. 2020;75(1):85-98. doi: 10.3233/JAD-191223. PMID 32280092
- [Background] Fan L, Zhu X, Sun S, Yu C, Huang X, Ness R, Dugan LL, Shu L, Seidner DL, Murff HJ, Fodor AA, Azcarate-Peril MA, Shrubsole MJ, Dai Q. Ca:Mg ratio, medium-chain fatty acids, and the gut microbiome. Clin Nutr. 2022 Nov;41(11):2490-2499. doi: 10.1016/j.clnu.2022.08.031. Epub 2022 Sep 12. PMID 36223712
- [Background] Fan L, Yu D, Zhu X, Huang X, Murff HJ, Azcarate-Peril MA, Shrubsole MJ, Dai Q. Magnesium and imidazole propionate. Clin Nutr ESPEN. 2021 Feb;41:436-438. doi: 10.1016/j.clnesp.2020.12.011. Epub 2021 Jan 7. PMID 33487303

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants, aged 40-85 y, with colorectal polyp or polyp-free individuals with high risk of colorectal cancer and had a calcium intake of ≥700 and <2000 mg/d, and their calcium-to-magnesium intake ratio was >2.6 (based on baseline two 24-hour dietary recalls) and have blood samples were recruited from Vanderbilt patient sources from March 11, 2011 to Jan 30, 2016 .
Period: Overall Study
Arm/Group | Magnesium Treatment | Placebo
Started | 124 | 126
Completed | 119 | 120
Not Completed | 5 | 6
Not completed — Withdrawal by Subject | 1 | 3
Not completed — Adverse Event | 4 | 2
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Magnesium Treatment | Placebo | Total
Number analyzed (Participants) | 119 | 120 | 239
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 82 | 78 | 160
  >=65 years | 37 | 42 | 79
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.1 (7.7) | 61.2 (8.1) | 60.7 (7.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 55 | 58 | 113
  Male | 64 | 62 | 126
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 1 | 3
  White | 117 | 119 | 236
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 119 | 120 | 239

OUTCOME MEASURES:

1. Primary Outcome: Changes of Cytosine Modification in TMPRSS2 (5-mC at cg16371860) by Magnesium Treatment Versus Placebo
Description: Increases in 5-mC methylation at cg16371860 (the promoter) indicate a hindered process of transcription initiation and, subsequently, lower levels of TMPRSS2 expression.
  5-mC methylation changes=value at 12 weeks minus value at baseline.
Time Frame: 12 Weeks
Population: Overall analysis and stratified analysis by age (<65 years, ≥ 65 years)
Measure: Mean (Standard Deviation); unit: units on CpG sites
Arm/Group | Magnesium Treatment | Placebo
Number analyzed (Participants) | 119 | 120
units on CpG sites
  All | 0.007 (0.024) | -0.001 (0.025)
  Age<65: number analyzed (Participants) | 82 | 78
  Age<65 | 0.012 (0.022) | -0.002 (0.022)
  Age≥65: number analyzed (Participants) | 37 | 42
  Age≥65 | -0.004 (0.025) | -0.001 (0.031)
Statistical Analysis 1: Comparison: Magnesium Treatment vs Placebo; Test type: Superiority; p < 0.05, Regression, Linear; P value was calculated using general linear model adjusted for age, sex, and baseline level

2. Secondary Outcome: Changes of Cytosine Modification in TMPRSS2 (5-hmC at cg16371860) by Magnesium Treatment Versus Placebo
Description: Decreases in 5-hmC methylation at cg16371860 (the promoter) indicate a hindered process of transcription initiation and, subsequently, lower levels of TMPRSS2 expression.
  5-hmC methylation changes=value at 12 weeks minus value at baseline.
Time Frame: 12 Weeks
Population: Overall analysis and stratified analysis by age (<65 years, ≥ 65 years)
Measure: Mean (Standard Deviation); unit: units on CpG sites
Arm/Group | Magnesium Treatment | Placebo
Number analyzed (Participants) | 119 | 120
units on CpG sites
  All | -0.001 (0.002) | 0.000 (0.002)
  Age<65: number analyzed (Participants) | 82 | 78
  Age<65 | -0.001 (0.002) | 0.000 (0.002)
  Age≥65: number analyzed (Participants) | 37 | 42
  Age≥65 | -0.000 (0.002) | 0.000 (0.002)
Statistical Analysis 1: Comparison: Magnesium Treatment vs Placebo; Test type: Superiority; p > 0.05, Regression, Linear; P value was calculated using general linear model adjusted for age, sex, and baseline level

3. Secondary Outcome: Changes of Cytosine Modification in TMPRSS2 (5-mC at cg26337277) by Magnesium Treatment Versus Placebo
Description: Increases in 5-mC methylation at cg26337277 (the promoter) indicate a hindered process of transcription initiation and, subsequently, lower levels of TMPRSS2 expression.
  5-mC methylation changes=value at 12 weeks minus value at baseline.
Time Frame: 12 Weeks
Population: Overall analysis and stratified analysis by age (<65 years, ≥ 65 years)
Measure: Mean (Standard Deviation); unit: units on CpG sites
Arm/Group | Magnesium Treatment | Placebo
Number analyzed (Participants) | 119 | 120
units on CpG sites
  All | 0.000 (0.001) | 0.000 (0.002)
  Age<65: number analyzed (Participants) | 82 | 78
  Age<65 | -0.000 (0.002) | -0.000 (0.002)
  Age≥65: number analyzed (Participants) | 37 | 42
  Age≥65 | 0.000 (0.001) | 0.000 (0.002)
Statistical Analysis 1: Comparison: Magnesium Treatment vs Placebo; Test type: Superiority; p > 0.05, Regression, Linear; P value was calculated using general linear model adjusted for age, sex, and baseline level

4. Secondary Outcome: Changes of Cytosine Modification in TMPRSS2 (5-hmC at cg26337277) by Magnesium Treatment Versus Placebo
Description: Decreases in 5-hmC methylation at cg26337277 (the promoter) indicate a hindered process of transcription initiation and, subsequently, lower levels of TMPRSS2 expression.
  5-hmC methylation changes=value at 12 weeks minus value at baseline.
Time Frame: 12 Weeks
Population: Overall analysis and stratified analysis by age (<65 years, ≥ 65 years)
Measure: Mean (Standard Deviation); unit: units on CpG sites
Arm/Group | Magnesium Treatment | Placebo
Number analyzed (Participants) | 119 | 120
units on CpG sites
  All | -0.000 (0.001) | 0.000 (0.001)
  Age<65: number analyzed (Participants) | 82 | 78
  Age<65 | -0.000 (0.001) | 0.000 (0.001)
  Age≥65: number analyzed (Participants) | 37 | 42
  Age≥65 | -0.000 (0.001) | 0.000 (0.001)
Statistical Analysis 1: Comparison: Magnesium Treatment vs Placebo; Test type: Superiority; p = 0.08, Regression, Linear; P value was calculated using general linear model adjusted for age, sex, and baseline level

ADVERSE EVENTS:
Time Frame: In the 12 weeks trial, we conducted safety and compliance calls to collect adverse event data.
Description: The definition of adverse event and/or serious adverse event is from the clinicaltrials.gov Definitions.
  We conducted safety and compliance calls to collect adverse event data.
Arm/Group | Magnesium Treatment | Placebo
All-Cause Mortality (participants affected / at risk) | 0/124 | 0/126
Serious Adverse Events (participants affected / at risk) | 0/124 | 0/126
Other Adverse Events (participants affected / at risk) | 4/124 | 3/126
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Magnesium Treatment (N=124) | Placebo (N=126)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 2 (2) — abdominal pain, stomach hurt
Bleeding after the rectal biopsy procedure (Gastrointestinal disorders) | 0 (0) | 1 (1)
Feel sick (General disorders) | 1 (1) | 0 (0)
Arthritic pain in fingers (General disorders) | 1 (1) | 0 (0)
Weight gain (General disorders) | 1 (1) | 0 (0) — 10 pound weight gain
Interaction with blood pressure medication (Vascular disorders) | 1 (1) | 0 (0) — may be having an adverse effect on blood pressure medication

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-06-08): https://cdn.clinicaltrials.gov/large-docs/03/NCT04196803/Prot_SAP_000.pdf